CLINICAL TRIAL: NCT02061813
Title: A 21-Day, Randomized, Controlled Study to Evaluate the Irritation Potential of Abametapir Lotion in Healthy Volunteers, Using a Cumulative Irritant Patch Test Design
Brief Title: Dermal Safety Study to Evaluate Potential Irritation of Abametapir Lotion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ha03-007
Record Dates: First submitted 2014-02-07; First posted 2014-02-13 (Estimated); Results first posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Head Lice
Keywords: Hatchtech
MeSH Terms: interventions — Sodium Dodecyl Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Abametapir lotion 0.74% w/w (Experimental): Applied 0.2 mL topically under occlusive condition
  Interventions: Drug: Abametapir Lotion 0.74% w/w
- Vehicle lotion (Placebo Comparator): Applied 0.2 mL topically under occlusive condition
  Interventions: Drug: Placebo
- Sodium Lauryl Sulfate (Other): Positive control applied 0.2 mL topically under occlusive condition
  Interventions: Drug: Sodium Lauryl Sulfate
- Saline 0.9% (Other): Negative control applied 0.2 mL topically under occlusive condition
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Abametapir Lotion 0.74% w/w — applied 0.2 mL topically under occlusive condition
  Arms: Abametapir lotion 0.74% w/w
Drug: Sodium Lauryl Sulfate — Sodium Lauryl Sulfate is prepared as a 0.2% aqueous solution by the site for topical administration, and applied 21 times over consecutive days under occlusive conditions, will serve as a positive control.
  Arms: Sodium Lauryl Sulfate
Drug: Saline 0.9% — A solution of 0.9% saline for topical administration, applied 21 times over consecutive days under occlusive conditions, will serve as a negative control
  Arms: Saline 0.9%
Drug: Placebo
  Arms: Vehicle lotion

SUMMARY:
The purpose of the study is to determine the irritation potential of repeat applications of abametapir lotion on normal skin.

DETAILED DESCRIPTION:
This will be a randomized, evaluator-blind, single-center, controlled, within-subject comparison study of the investigational products (abametapir lotion) and its vehicle lotion and positive and negative controls under occlusive conditions in healthy volunteers. All subjects will have the investigational product (abametapir lotion), the vehicle product, the positive control patch, and negative control patch applied to 4 randomly assigned, adjacent skin sites on the infrascapular area of their back, for the purpose of determining irritation potential.

The investigational products, vehicle, and controls will be applied to one side of the infrascapular area of the back. Evaluation of dermal reactions at the application sites will be assessed clinically using a visual scale that rates the degree of erythema, edema, and other signs of cutaneous irritation (see Section 3.5.5).

A total of 21 applications of each product will be made.

ELIGIBILITY:
Inclusion Criteria:

1. Are healthy (to be confirmed by medical history) males or females, 18 years of age or older;
2. In the case of females of childbearing potential, are using an acceptable form of birth control (oral/implant/injectable/transdermal contraceptives, intrauterine device, condom with spermicide, diaphragm with spermicide, abstinence, partner's vasectomy). Abstinence or vasectomized partner are acceptable if the female subject agrees to implement one of the other acceptable methods of birth control if her lifestyle/partner changes;
3. If female of childbearing potential, have a negative urine pregnancy test (UPT) at Day 1, and are willing to submit to a pregnancy test at the end of study (EOS);
4. Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events;
5. Are of any skin type or race, providing the skin pigmentation will allow discernment of erythema;
6. Complete a patch study Medical Screening form as well as a Medical Personal History form; and
7. Read, understand, and provide signed informed consent.

Exclusion Criteria:

1. Have any visible skin disease at the application site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test site reaction;
2. Are not willing to refrain from using topical/systemic analgesics such as aspirin (daily use of 81 mg aspirin is acceptable), Aleve, Motrin, Advil, or Nuprin for 72 hours prior to and during the study (occasional use of acetaminophen will be permitted);
3. Are using inhaled/systemic/topical corticosteroids in the 3 weeks prior to and during the study, or systemic/topical antihistamines for 72 hours prior to and during the study;
4. Are using medication which, in the opinion of the investigative personnel, will interfere with the study results, including anti-inflammatory medications;
5. Are unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions, or similar products on the back during the study;
6. Have psoriasis and/or active atopic dermatitis/eczema;
7. Are females who are pregnant, plan to become pregnant during the study, or are breast-feeding a child;
8. Have a known sensitivity to constituents present in the material being evaluated;
9. Have damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site
10. Have received treatment for any type of internal cancer within 5 years prior to study entry;
11. Have a history of, or are currently being treated for skin cancer;
12. Are currently participating in any other clinical trial,
13. Have any known sensitivity to adhesives; and/or
14. Have received any investigational treatment(s) within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dosik, Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Reserach Inc, Paramus, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Skin sites
Groups:
- All Randomized Subjects: All Randomized Subjects included all subjects who were enrolled into the study. All subjects had the investigational product (abametapir lotion), the vehicle product, the positive control patch, and negative control patch applied to 4 randomly assigned, adjacent skin sites on the infrascapular area of their back, for the purpose of determining irritation potential.
Period: Overall Study
Arm/Group | All Randomized Subjects
Started | 40; 160 Skin sites
Abametapir Lotion | 40; 40 Skin sites
Vehicle Lotion | 40; 40 Skin sites
Saline 0.9% | 40; 40 Skin sites
SLS 0.2% | 40; 40 Skin sites
Completed | 37; 148 Skin sites
Not Completed | 3; 12 Skin sites
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | All Randomized Subjects
Number analyzed (Participants) | 40
Age, Customized [Mean (Standard Deviation); unit: years] | 46.95 (14.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick (FP) Scale is a numerical classification schema for human skin color. FP 1 is for white skin type and progressively becoming darker until FP 6 which is for black skin type.
  FP 1 = Always burns easily, never tans; FP 2 = Always burns easily, tans minimally; FP 3 = Burns moderately, tans gradually (light brown); FP 4 = Burns minimally, always tans well (moderate brown); FP 5 = Rarely burns, tans very well (moderate brown); FP 6 = Never burns, deeply pigmented
  Participants
    Fitzpatrick Type 1 | 1
    Fitzpatrick Type 2 | 15
    Fitzpatrick Type 3 | 11
    Fitzpatrick Type 4 | 12
    Fitzpatrick Type 5 | 1

OUTCOME MEASURES:

1. Primary Outcome: Potential of Abametapir Lotion to Cause Irritation After Repeated Topical Application to the Healthy Skin of Humans.
Description: The evaluation of irritation is based on Modified Berger procedure and is accepted as standard methodology for assessment of cumulative irritation potential. The assessment of all patch sites for irritation symptoms will be visually assessed by a trained evaluator using the numerical equivalents (0-7) where 0 is the least irritation potential and 7 is the maximum irritation potential. The scoring will be done on daily basis from baseline through Day 21 visit. The final reported outcome is a mean of the scores over 21 days.
Time Frame: 21 days
Population: All Randomized Subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Skin Sites
Groups:
- Abametapir Lotion Group; Vehicle Lotion; Saline 0.9%; Sodium Lauryl Sulphate (SLS): All Subjects in the study received all treatments simultaneously on a daily basis, as it was an intra-subject comparison design
Arm/Group | Abametapir Lotion Group | Vehicle Lotion | Saline 0.9% | Sodium Lauryl Sulphate (SLS)
Number analyzed (Participants) | 40 | 40 | 40 | 40
Number analyzed (Skin Sites) | 40 | 40 | 40 | 40
score on a scale | 1.10 (3.11) | 0.70 (2.89) | 1.10 (6.48) | 49.15 (8.87)

ADVERSE EVENTS:
Time Frame: All Adverse events were systematically recorded from the time of signing informed consent until the last assessment i.e. 21 days.
Groups:
- All Randomized Subjects: All Randomized Subjects included all subjects who were enrolled into the study. All subjects received application of all four interventions.
Arm/Group | All Randomized Subjects
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No